CLINICAL TRIAL: NCT01089972
Title: Ultrasonographic Evaluation of the Radial and Ulnar Blood Flow After Radial Arterial Cannulation
Status: Completed | Type: Observational
Sponsor: Severance Hospital (Other)
Responsible Party: Severance Hospital, Anesthesia and Pain Research Institute
Other Study IDs: IRB 1-2009-0033
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2010-03

CONDITIONS: Radial Artery, Regional Blood Flow
Keywords: radial artery; ulnar artery; catheterization; regional blood flow

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 20 gauge group
  Interventions: Device: 20 gauge catheter
- 22 gauge group
  Interventions: Device: 22 gauge catheter

INTERVENTIONS:
Device: 22 gauge catheter — radial artery cannulation using 22 gauge catheter
  Groups: 22 gauge group
Device: 20 gauge catheter — radial artery cannulation using 20 gauge catheter
  Groups: 20 gauge group

SUMMARY:
The aim of this randomized study was to compare the impact of two different radial arterial catheters - 20G and 22G - on the changes of diameter, blood flow and velocity of radial artery and ulnar artery after induction of anesthesia and after cannulation.

ELIGIBILITY:
Inclusion Criteria:

* The patient who are scheduled for elective surgery and need arterial cannulation

Exclusion Criteria:

* Coronary occlusive disease
* Known or suspected upper extremity peripheral arterial disease
* Coagulopathy
* DM with peripheral neuropathy
* Infection at puncture site

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient(age >20) who are scheduled for elective surgery and need arterial
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Radial artery diameter and blood flow before and after cannulation | 30 min
Ulnar artery diameter and blood flow before and after cannulation | 30 min

SECONDARY OUTCOMES:
The differences of radial artery diameter and blood flow after cannulation between catheter gauge(20- and 22-G) | 30 min
The differences of ulnar artery diameter and blood flow after cannulation between catheter gauge(20- and 22-G) | 30 min

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea